CLINICAL TRIAL: NCT04027348
Title: Palliative Management of Inoperable Malignant Bowel Obstruction: A Prospective, Open Label, Phase-2 Study at an NCI Comprehensive Cancer Center
Brief Title: Palliative Management of Inoperable Malignant Bowel Obstruction
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 74018
Record Dates: First submitted 2019-07-18; First posted 2019-07-22 (Actual); Results first posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-09

CONDITIONS: Malignant Bowel Obstruction
Keywords: bowel obstruction
MeSH Terms: conditions — Intestinal Obstruction | interventions — Dexamethasone; Metoclopramide; Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (octreotide, dexamethasone, metoclopramide) (Experimental): IV octreotide 300 mcg TID + IV dexamethasone 4 mg BID (first dose 9am and second at 2pm) + IV metoclopramide 10 mg q6h.
  Interventions: Drug: Dexamethasone; Drug: Metoclopramide; Drug: Octreotide

INTERVENTIONS:
Drug: Dexamethasone — Given IV
Drug: Metoclopramide — Given IV
Drug: Octreotide — Given IV

SUMMARY:
To identify the role of palliative medical management of inoperable malignant bowel obstruction (MBO) with Octreotide, Dexamethasone and Metoclopramide given together as triple therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age.
* Diagnosis of partial bowel obstruction secondary to active or prior malignancy (primary or metastatic GI, GYN, and carcinomatosis) caused either by tumor itself or adhesions inthe setting of active malignancy.
* Cross-sectional imaging performed within 24 hours of clinical symptoms of bowel obstruction (nausea, vomiting, and constipation ± abdominal pain) during hospital admission.
* Patient must have an inoperable MBO
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved writteninformed consent form prior to receiving any study related procedure.

Exclusion Criteria:

* Evidence of complete bowel obstruction by imaging.
* Bacteremia/septicemia with a documented positive blood culture: If a blood culture comes back positive after study enrollment, patient will be excluded.
* Patients already taking a steroid equivalent to 8 mg of dexamethasone per day prior to study enrollment.
* Patients undergoing bowel surgery or stent placement for bowel obstruction.
* Those patients with MBO in setting of incarcerated hernia.
* Known history of QT prolongation syndrome or if QTc is > 450 msec in males or > 470 msec in females on baseline EKG within 2 weeks of enrollment.
* Lack of decision making capacity/delirium.
* Pregnant or nursing female participants.
* Actively suicidal patients.
* Acute cholecystitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Case, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Octreotide, Dexamethasone, Metoclopramide)
Started | 15
Completed | 13
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Octreotide, Dexamethasone, Metoclopramide)
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 15
Performance Status [Mean (Standard Deviation); unit: units on a scale] — KARNOFSKY PERFORMANCE STATUS SCALE
  The Karnofsky Performance Scale Index allows patients to be classified as to their functional impairment. This can be used to compare effectiveness of different therapies and to assess the prognosis in individual patients. The lower the Karnofsky score, the worse the survival for most serious illnesses.
  The score ranges from 0 to 100.
  units on a scale | 64.7 (18.9)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Obstruction Clearance
Description: The primary efficacy endpoint is the proportion of eligible patients whose malignant bowel obstruction clears (de-obstruction) within 7 days of starting the protocol therapy. Patients meeting de-obstruction criteria within 7 days will be deemed treatment successes.
  De-obstruction is defined as:
  * Effective introduction of oral intake (yes/no)
  * Distinguished from small volumes of oral fluid that may be allowed with unresolved MBO
  * Tolerating oral liquid diet (day 1 of de-obstruction) that is able to be progressively more solid (oral or enteral)
  * Cessation of vomiting or ability for NGT or venting G tube to remain clamped without vomiting
  Rate of de-obstruction is defined as:
  - From the date of study enrollment to the first observation of de-obstruction.
Time Frame: Within 7 days of starting protocol therapy
Population: 2 Patients did not complete treatment and were not evaluated for de-obstruction (due to AEs).
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Octreotide, Dexamethasone, Metoclopramide)
Number analyzed (Participants) | 13
Participants | 10

ADVERSE EVENTS:
Time Frame: From start of treatment up to 30-days after treatment, where treatment was an average of 2 weeks.
Arm/Group | Treatment (Octreotide, Dexamethasone, Metoclopramide)
All-Cause Mortality (participants affected / at risk) | 13/15
Serious Adverse Events (participants affected / at risk) | 6/15
Other Adverse Events (participants affected / at risk) | 11/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Octreotide, Dexamethasone, Metoclopramide) (N=15)
Obstruction gastric (Gastrointestinal disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Octreotide, Dexamethasone, Metoclopramide) (N=15)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 5 (6)
Vomiting (Gastrointestinal disorders) | 2 (2)
Edema limbs (General disorders) | 3 (3)
Fatigue (General disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Thrush (Infections and infestations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 4 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-21): https://cdn.clinicaltrials.gov/large-docs/48/NCT04027348/Prot_SAP_000.pdf